CLINICAL TRIAL: NCT01522144
Title: EHR Decision Support to Improve Outpatient Asthma Care
Brief Title: An Electronic Decision Support Tool to Improve Outpatient Asthma Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, lbell, Medical Director of PeRC, Agency for Healthcare Research and Quality (AHRQ)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: R21HS014873 (AHRQ)
Record Dates: First submitted 2012-01-19; First posted 2012-01-31 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Electronic Health Records

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Asthma clinical decision support (Experimental): decision support compared to no decision support in a cluster-randomized trial by practise
  Interventions: Behavioral: Computerized Decision support

INTERVENTIONS:
Behavioral: Computerized Decision support — Using a clustered randomized method, computerized decision support, embedded in the electronic health record, was offered to selected primary care practices and outcomes of asthma care were compared to those practices without the computerized decision support.
  Other Names: electronic health record

SUMMARY:
The Children's Hospital of Philadelphia's ambulatory network uses an electronic health record (EHR) to document clinical information. Using the EHR, a clinical decision support tool will be designed to help the primary care physician's in caring for children with asthma. The goal will be to improve the primary care physician's use of the national Institutes of Health guidelines for the best care for asthma. To study this EHR decision support tool, it will be introduced into 5 practices while 5 other practices will have the existing asthma care information. It will be determined whether the physicians in the practices with the decision support tool are better at following the asthma guidelines. If the decision support tool works...then it will be offered to others to use with their EHR systems.

DETAILED DESCRIPTION:
National Asthma Education and Prevention Program guidelines (NAEPP) exist, but are under used in Primary Care. In addition, implementation of the guidelines has been shown to be vary according to the location of practice and other contextual factors.

The Children's Hospital of Philadelphia Pediatric Research Consortium (PeRC), a practice-based research network will determine whether an innovative clinical decision support system embedded in an existing electronic health record (EHR) will improve provider adherence to the existing NAEPP guidelines.

After receiving a standardized education module based on NAEPP guidelines, 10 primary care pediatric practices (both urban and suburban) will be randomized to receive either a passive EHR (control sites) or an interactive decision support sytem (intervention sites).

The primary outcome of interest will be the proportion of patient son appropriate asthma controller medication compared over time. Secondary outcomes include the proportion of asthma patients with: 1) an updated asthma action plan 2) documentation of spirometry performed (6 to 17years) and 3) an updated problem list reflecting current asthma severity. After hours calls to providers and types of office visits related to to asthma will be tracked. Contextual factors at the clinic and patient level will be examined to assess their association with the outcomes of interest. In addition, measurement of asthma-related quality of life and missed school and work in a sample of 200 subjects from each group will be performed

If shown to be successful, this type of clinical decision support, embedded within the EHR, has the potential to be a powerful tool to improve the implementation of asthma guidelines and clinical practice guidelines for other conditions and illnesses.

ELIGIBILITY:
Inclusion Criteria:

* Children with the diagnosis of asthma
* Children enrolled in one of 10 selected primary care practices in the PeRC practice-based research network

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1030 (Actual)
Dates: Start 2006-07; Primary Completion 2008-04 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
The proportion of patients on appropriate asthma controller medication at the end of the trial | assessed at each visit
  each patient who is classified as having persistant asthma should be on at least one appropriate controller medication for asthma.

SECONDARY OUTCOMES:
1) an updated asthma action plan | updated at least once per year
  Each patient should have an asthma care plan updated once per year
2)documentation of spirometry(6 to 18 yrs)in those with asthma | spirometry should be done once per year
  Each patient should have had spirometry at least once per year.
3) an updated problem list that reflects an assessment of asthma severity | tthe asthma severity should be on the problem list
  each patient should have their asthma severity classification on the thier chart

CONTACTS AND LOCATIONS:
Overall Officials: Louis M Bell, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Asthma mortality and hospitalization among children and young adults--United States, 1980-1993. From the Centers for Disease Control and Prevention. JAMA. 1996 May 22-29;275(20):1535-7. No abstract available. PMID 8622235
- [Background] Lieu TA, Quesenberry CP Jr, Capra AM, Sorel ME, Martin KE, Mendoza GR. Outpatient management practices associated with reduced risk of pediatric asthma hospitalization and emergency department visits. Pediatrics. 1997 Sep;100(3 Pt 1):334-41. doi: 10.1542/peds.100.3.334. PMID 9282702
- [Background] Landry P, Tremblay S, Darioli R, Genton B. Inactivated hepatitis A vaccine booster given >/=24 months after the primary dose. Vaccine. 2000 Oct 15;19(4-5):399-402. doi: 10.1016/s0264-410x(00)00188-2. PMID 11027799